CLINICAL TRIAL: NCT05719220
Title: The Effect of Group Preoperative Pelvic Floor Training on Transient Urinary Incontinence After Holmium Laser Enucleation of the Prostate: A Prospective Cohort Study
Brief Title: Effect of Group Preoperative Pelvic Floor Training for HoLEP
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 23-38400
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: BPH; Urinary Incontinence
Keywords: benign prostatic hyperplasia; pelvic floor training; group therapy; holmium laser enucleation of the prostate; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group preoperative pelvic floor training: Patients will receive group preoperative PFT, 4 weeks prior to HoLEP.
  Interventions: Behavioral: Group preoperative pelvic floor training
- No preoperative pelvic floor training: The control group will receive standard care, which may include patient education about postoperative care and pelvic floor muscle exercises, but will not receive structured group PFT.

INTERVENTIONS:
Behavioral: Group preoperative pelvic floor training — Patients will receive PFT from a trained physical therapist delivered in a group setting of 8-10 people. The investigators allow patients in the PFT group to attend group classes as many times as they want prior to surgery to see if the frequency of training has an effect on outcomes. The treatment group could be required to go to at least 1 group class 4 weeks prior to their procedure, but they could be welcome to attend more if they want further practice and review of the material. A 45-minute group class with basic PFT guidelines could be presented weekly during the study.
  Groups: Group preoperative pelvic floor training

SUMMARY:
The main goal of this study is to see if group pelvic floor training before surgery can help prevent urinary incontinence after Holmium laser enucleation of the prostate (HoLEP) surgery. The study has the potential to inform preoperative intervention strategies for managing incontinence after HoLEP.

DETAILED DESCRIPTION:
Preoperative pelvic floor training (PFT) may improve early urinary incontinence after prostate surgery. Group-based training potentially provides additional benefits such as cost-benefit, social support, and motivation. However, the efficacy of group preoperative PFT has not been reported. This study aims to determine the effect of group preoperative PFT on transient urinary incontinence after HoLEP in a prospective cohort of patients and to identify any potential predictors of transient urinary incontinence after HoLEP.

In this study, the investigators will recruit approximately 50 patients in each cohort (total 100) and will be followed over time to collect data on both the exposure (group PFT) and the outcome (incidence of urinary incontinence 1 month and 3 months after HoLEP). Potential confounding variables, such as patient demographics, preoperative imaging, and operative data, will be collected and analyzed. The results of this study have the potential to inform the development of effective preoperative interventions for the management of transient urinary incontinence after HoLEP.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a diagnosis of BPH with a plan to undergo HoLEP.
* Between the age of 50-90.
* Ability to understand and provide informed consent.

Exclusion Criteria:

* Patients whom inability to carry out PFT protocol.
* Patients unwilling or unable to complete follow up care.
* Severe urinary incontinence due to a history of neurological diseases such as a cerebrovascular accident or spinal cord injuries.
* Patients whom inability to read and understand the English language.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit a cohort of patients scheduled to undergo HoLEP at the UCSF Urology Clinic. Well-informed consent will be obtained from every patient after giving balanced information about the options of group preoperative PFT and no training before recruitment in the study. The investigators will offer the group class to everyone and use the patients who decline the group class as the control group (N = 50: 50 each arm).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of urinary incontinence at 1 month | 1 month after the operation
  Urinary incontinence (present/absent) will be defined according to the guidelines of the International Continence Society as involuntary loss of urine experienced during the bladder storage phase using self-report measures at regular intervals postoperatively.
Incidence of urinary incontinence at 3 months | 3 months after the operation
  Urinary incontinence (present/absent) will be defined according to the guidelines of the International Continence Society as involuntary loss of urine experienced during the bladder storage phase using self-report measures at regular intervals postoperatively.

SECONDARY OUTCOMES:
The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form at 1 month | 1 month after the operation
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a self-administered questionnaire used to measure the severity of urinary incontinence symptoms, such as frequency, urgency, and amount of urine loss, as well as the impact of urinary incontinence on daily activities and emotional well-being. The total score ranges from 0 to 21, with higher scores indicating more severe urinary incontinence and greater impact on quality of life.
The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form at 3 months | 3 months after the operation
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a self-administered questionnaire used to measure the severity of urinary incontinence symptoms, such as frequency, urgency, and amount of urine loss, as well as the impact of urinary incontinence on daily activities and emotional well-being. The total score ranges from 0 to 21, with higher scores indicating more severe urinary incontinence and greater impact on quality of life.
The International Prostate Symptom Score at 1 month | 1 month after the operation
  The International Prostate Symptom Score (IPSS) is a self-administered questionnaire that assesses the severity of lower urinary tract symptoms (LUTS) in men. The questionnaire consists of 7 items that assess symptoms such as frequency, urgency, nocturia, weak stream, straining, incomplete emptying, and terminal dribbling. Each item is scored on a scale of 0-5. The total score ranges from 0 to 35, with higher scores indicating more severe symptoms and the last question for measuring the effect of LUTS on quality of life.
The International Prostate Symptom Score at 3 months | 3 months after the operation
  The International Prostate Symptom Score (IPSS) is a self-administered questionnaire that assesses the severity of lower urinary tract symptoms (LUTS) in men. The questionnaire consists of 7 items that assess symptoms such as frequency, urgency, nocturia, weak stream, straining, incomplete emptying, and terminal dribbling. Each item is scored on a scale of 0-5. The total score ranges from 0 to 35, with higher scores indicating more severe symptoms and the last question for measuring the effect of LUTS on quality of life.
Pelvic floor muscle strength at 1 month | 1 month after the operation
  Preoperative and postoperative pelvic floor muscle strength measured by perineometer (the output in cmH2O) will be compared to determine whether the strength gain or maintenance, which could be a repeated measure at baseline, 1 month, and 3 months.
Pelvic floor muscle strength at 3 months | 3 months after the operation
  Preoperative and postoperative pelvic floor muscle strength measured by perineometer (the output in cmH2O) will be compared to determine whether the strength gain or maintenance, which could be a repeated measure at baseline, 1 month, and 3 months.
Patient satisfaction | Immediately after the completion of the PFT program or soon thereafter
  Patient satisfaction after receiving group PFT will be evaluated using a patient satisfaction with outpatient physical therapy survey.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilling PJ, Wilson LC, King CJ, Westenberg AM, Frampton CM, Fraundorfer MR. Long-term results of a randomized trial comparing holmium laser enucleation of the prostate and transurethral resection of the prostate: results at 7 years. BJU Int. 2012 Feb;109(3):408-11. doi: 10.1111/j.1464-410X.2011.10359.x. Epub 2011 Aug 23. PMID 21883820
- [Background] Sun F, Sun X, Shi Q, Zhai Y. Transurethral procedures in the treatment of benign prostatic hyperplasia: A systematic review and meta-analysis of effectiveness and complications. Medicine (Baltimore). 2018 Dec;97(51):e13360. doi: 10.1097/MD.0000000000013360. PMID 30572440
- [Background] Lerner LB, McVary KT, Barry MJ, Bixler BR, Dahm P, Das AK, Gandhi MC, Kaplan SA, Kohler TS, Martin L, Parsons JK, Roehrborn CG, Stoffel JT, Welliver C, Wilt TJ. Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: AUA GUIDELINE PART II-Surgical Evaluation and Treatment. J Urol. 2021 Oct;206(4):818-826. doi: 10.1097/JU.0000000000002184. Epub 2021 Aug 13. PMID 34384236
- [Background] Cho MC, Park JH, Jeong MS, Yi JS, Ku JH, Oh SJ, Kim SW, Paick JS. Predictor of de novo urinary incontinence following holmium laser enucleation of the prostate. Neurourol Urodyn. 2011 Sep;30(7):1343-9. doi: 10.1002/nau.21050. Epub 2011 Apr 28. PMID 21538499
- [Background] Nam JK, Kim HW, Lee DH, Han JY, Lee JZ, Park SW. Risk Factors for Transient Urinary Incontinence after Holmium Laser Enucleation of the Prostate. World J Mens Health. 2015 Aug;33(2):88-94. doi: 10.5534/wjmh.2015.33.2.88. Epub 2015 Aug 19. PMID 26331125
- [Background] Shigemura K, Tanaka K, Yamamichi F, Chiba K, Fujisawa M. Comparison of Predictive Factors for Postoperative Incontinence of Holmium Laser Enucleation of the Prostate by the Surgeons' Experience During Learning Curve. Int Neurourol J. 2016 Mar;20(1):59-68. doi: 10.5213/inj.1630396.198. Epub 2016 Mar 9. PMID 27032559
- [Background] Houssin V, Olivier J, Brenier M, Pierache A, Laniado M, Mouton M, Theveniaud PE, Baumert H, Mallet R, Marquette T, Villers A, Robert G, Rizk J. Predictive factors of urinary incontinence after holmium laser enucleation of the prostate: a multicentric evaluation. World J Urol. 2021 Jan;39(1):143-148. doi: 10.1007/s00345-020-03169-0. Epub 2020 Mar 26. PMID 32219512
- [Background] Pan LH, Lin MH, Pang ST, Wang J, Shih WM. Improvement of Urinary Incontinence, Life Impact, and Depression and Anxiety With Modified Pelvic Floor Muscle Training After Radical Prostatectomy. Am J Mens Health. 2019 May-Jun;13(3):1557988319851618. doi: 10.1177/1557988319851618. PMID 31092098
- [Background] MacDonald R, Fink HA, Huckabay C, Monga M, Wilt TJ. Pelvic floor muscle training to improve urinary incontinence after radical prostatectomy: a systematic review of effectiveness. BJU Int. 2007 Jul;100(1):76-81. doi: 10.1111/j.1464-410X.2007.06913.x. Epub 2007 Apr 13. PMID 17433028
- [Background] Centemero A, Rigatti L, Giraudo D, Lazzeri M, Lughezzani G, Zugna D, Montorsi F, Rigatti P, Guazzoni G. Preoperative pelvic floor muscle exercise for early continence after radical prostatectomy: a randomised controlled study. Eur Urol. 2010 Jun;57(6):1039-43. doi: 10.1016/j.eururo.2010.02.028. Epub 2010 Mar 1. PMID 20227168
- [Background] Chang JI, Lam V, Patel MI. Preoperative Pelvic Floor Muscle Exercise and Postprostatectomy Incontinence: A Systematic Review and Meta-analysis. Eur Urol. 2016 Mar;69(3):460-7. doi: 10.1016/j.eururo.2015.11.004. Epub 2015 Nov 21. PMID 26610857
- [Background] Anan G, Kaiho Y, Iwamura H, Ito J, Kohada Y, Mikami J, Sato M. Preoperative pelvic floor muscle exercise for early continence after holmium laser enucleation of the prostate: a randomized controlled study. BMC Urol. 2020 Jan 23;20(1):3. doi: 10.1186/s12894-019-0570-5. PMID 31973706
- [Background] Dumoulin C, Morin M, Danieli C, Cacciari L, Mayrand MH, Tousignant M, Abrahamowicz M; Urinary Incontinence and Aging Study Group. Group-Based vs Individual Pelvic Floor Muscle Training to Treat Urinary Incontinence in Older Women: A Randomized Clinical Trial. JAMA Intern Med. 2020 Oct 1;180(10):1284-1293. doi: 10.1001/jamainternmed.2020.2993. PMID 32744599
- [Background] Pereira VS, Correia GN, Driusso P. Individual and group pelvic floor muscle training versus no treatment in female stress urinary incontinence: a randomized controlled pilot study. Eur J Obstet Gynecol Reprod Biol. 2011 Dec;159(2):465-71. doi: 10.1016/j.ejogrb.2011.09.003. Epub 2011 Oct 1. PMID 21962461
- [Background] Lamb SE, Pepper J, Lall R, Jorstad-Stein EC, Clark MD, Hill L, Fereday-Smith J. Group treatments for sensitive health care problems: a randomised controlled trial of group versus individual physiotherapy sessions for female urinary incontinence. BMC Womens Health. 2009 Sep 14;9:26. doi: 10.1186/1472-6874-9-26. PMID 19751517
- [Background] D'Ancona C, Haylen B, Oelke M, Abranches-Monteiro L, Arnold E, Goldman H, Hamid R, Homma Y, Marcelissen T, Rademakers K, Schizas A, Singla A, Soto I, Tse V, de Wachter S, Herschorn S; Standardisation Steering Committee ICS and the ICS Working Group on Terminology for Male Lower Urinary Tract & Pelvic Floor Symptoms and Dysfunction. The International Continence Society (ICS) report on the terminology for adult male lower urinary tract and pelvic floor symptoms and dysfunction. Neurourol Urodyn. 2019 Feb;38(2):433-477. doi: 10.1002/nau.23897. Epub 2019 Jan 25. PMID 30681183
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Barry MJ. Evaluation of symptoms and quality of life in men with benign prostatic hyperplasia. Urology. 2001 Dec;58(6 Suppl 1):25-32; discussion 32. doi: 10.1016/s0090-4295(01)01300-0. PMID 11750246
- [Background] Beattie PF, Pinto MB, Nelson MK, Nelson R. Patient satisfaction with outpatient physical therapy: instrument validation. Phys Ther. 2002 Jun;82(6):557-65. PMID 12036397